CLINICAL TRIAL: NCT04195074
Title: Study on Therapeutic Effects and Safety of Three Types of Nucleotide/Nucleoside Analogues in Patients With Chronic Hepatitis b
Brief Title: Three Types of Nucleotide/Nucleoside Analogues Therapy in Patients With Chronic Hepatitis b
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL8
Record Dates: First submitted 2019-12-05; First posted 2019-12-11 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis b; nucleoside; nucleotide
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ETV group (Experimental): 100 patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day from baseline to life-long.
  Interventions: Drug: Entecavir
- TDF group (Experimental): 100 patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- TAF group (Experimental): 100 patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Entecavir — Patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day.
  Other Names: Baraclude
  Arms: ETV group
Drug: Tenofovir Disoproxil Fumarate — Patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day.
  Other Names: Viread
  Arms: TDF group
Drug: Tenofovir Alafenamide — Patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day.
  Other Names: Vemlidy
  Arms: TAF group

SUMMARY:
This study is to investigate the clinical efficacy and safety of three types of nucleotide/nucleoside analogues in treatment of chronic hepatitis b

DETAILED DESCRIPTION:
Chronic hepatitis b (CHB) remains a serious public health problem in China. Nucleotide/nucleoside analogues are used for anti-virus treatment in these patients. Entecavir, Tenofovir Disoproxil Fumarate and Tenofovir Alafenamide are first line drug in China. But there still lacks of data of Tenofovir Alafenamide in treatment of CHB. This study is to investigate the clinical efficacy and safety of three types of nucleotide/nucleoside analogues in treatment of CHB.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Age from 18 to 65 years old;
3. HBeAg-positive: HBV DNA≥20000IU/ml，HBeAg-negative: HBV DNA≥2000IU/ml；
4. ALT≥2×ULN；
5. Do not receive nucleotide/nucleoside analogues treatment in the past half year.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions;
7. Using glucocorticoid;
8. Patients can not follow-up;
9. Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of renal function decline | 144 week
  Renal function indicators mainly include blood urea nitrogen, serum creatine and estimated glomerular filtration rate, and the rate of renal function decline would be evaluated.
Rate of hypercalcemia | 144 week
  The serum calcium would be detected to know the ratio of patients with hypercalcemia.

SECONDARY OUTCOMES:
hepatitis b virus(HBV) DNA undetectable rate | 0 week, 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b virus DNA would not be detected if it below the upper limit of test value.
hepatitis b e antigen loss rate | 0 week, 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b e antigen would be tested to know the ratio of patients with negative hepatitis B e antigen.
hepatitis b s antigen loss rate | 0 week, 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b s antigen become negative and quantitative analysis below the upper limit of test value.
hepatitis b e antigen seroconversion rate | 0 week, 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  hepatitis b e antibody would be tested to know the ratio of patients with positive hepatitis B e antibody

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China